CLINICAL TRIAL: NCT06291038
Title: Efficacy of Glutamine Supplementation in Patients Suffering From Irritable Bowel
Brief Title: Efficacy of Glutamine Supplementation in Patients Suffering From Irritable Bowel Syndrome With Impaired Intestinal Permeability
Acronym: MISSISIIPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/0381/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Multicentric; prospective; randomized; double blind; interregional
Who Masked: Participant
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine (Experimental): • Experimental group: treatment with glutamine at a dose of 5g 3 times a day for 8 weeks.
  Interventions: Dietary Supplement: • Experimental group: treatment with glutamine at a dose of 5g 3 times a day for 8 weeks
- Protifar (Placebo Comparator): • Control group: treatment with a protein powder (Protifar) (Placébo) 5g 3 times a day for 8 weeks.
  Interventions: Dietary Supplement: • Control group: treatment with a protein powder (Protifar) (Placébo) 5g 3 times a day for 8 weeks.

INTERVENTIONS:
Dietary Supplement: • Experimental group: treatment with glutamine at a dose of 5g 3 times a day for 8 weeks — treatment with glutamine at a dose of 5g 3 times a day for 8 weeks
  Arms: Glutamine
Dietary Supplement: • Control group: treatment with a protein powder (Protifar) (Placébo) 5g 3 times a day for 8 weeks. — treatment with a protein powder (Protifar) (Placébo) 5g 3 times a day for 8 weeks.
  Arms: Protifar

SUMMARY:
Irritable bowel syndrome (IBS) affects approximately 5% of the general population and remains a daily problem in the practice of clinicians with inconsistent effectiveness of treatments while patients' expectations are high.

One of the functional abnormalities described during IBS is increased intestinal permeability. This increase in intestinal permeability is primarily present in the diarrheal subtype (IBS-D) and can be measured using the lactulose/mannitol test.

Glutamine is a non-essential amino acid which regulates numerous metabolic pathways, and which plays a key role in the intestine because it is the preferential substrate of enterocytes and immune cells. Ex vivo, glutamine is able to restore the expression of tight junction proteins in patients suffering from IBS-D. On the other hand, glutamine supplementation is capable of reducing abdominal pain and restoring intestinal permeability disorders in a subgroup of patients with intestinal permeability disorder (post-infectious IBS-D).

Our working hypothesis would be that all patients suffering from IBS with permeability disorder, measured by the lactulose/mannitol test, could benefit from oral glutamine supplementation.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) affects approximately 5% of the general population and remains a daily problem in the practice of clinicians with inconsistent effectiveness of treatments while patients' expectations are high.

One of the functional abnormalities described during IBS is increased intestinal permeability. This increase in intestinal permeability is primarily present in the diarrheal subtype (IBS-D) and can be measured using the lactulose/mannitol test.

Glutamine is a non-essential amino acid which regulates numerous metabolic pathways, and which plays a key role in the intestine because it is the preferential substrate of enterocytes and immune cells. Ex vivo, glutamine is able to restore the expression of tight junction proteins in patients suffering from IBS-D. On the other hand, glutamine supplementation is capable of reducing abdominal pain and restoring intestinal permeability disorders in a subgroup of patients with intestinal permeability disorder (post-infectious IBS-D).

Our working hypothesis would be that all patients suffering from IBS with permeability disorder, measured by the lactulose/mannitol test, could benefit from oral glutamine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 to 75
* Diarrheal irritable bowel syndrome (IBS-D), according to the Rome IV criteria (appendix 2)
* Francis score > 175/500 at inclusion (corresponding to moderate to severe IBS)
* Treatments for IBS stable for >1 month
* Affiliation to a social security system
* Adult person having read and understood the information letter and signed the consent form
* Woman of childbearing age having effective/very effective contraception (Cf. CTFG) (estrogen-progestins or intrauterine device or tubal ligation) for 1 month and a negative urine pregnancy test
* Postmenopausal woman: confirmatory diagnosis (amenorrhea not medically induced for at least 12 months before the inclusion visit or biologically documented)

Exclusion Criteria:

* Taking probiotics, anti-inflammatories, corticosteroids or antibiotics systemically (oral or injectable) in the month preceding the study and during the duration of the study treatment,
* Known diagnosis of active autoimmune disease (type 1 diabetes, lupus, multiple sclerosis, thyroiditis, ankylosing spondylitis, rheumatoid arthritis or psoriasis)
* Known allergy to glutamine,
* Contraindication to taking glutamine, protein powder, lactulose or mannitol (including sugar-free chewing gum),
* Use of osmotic laxatives and/or taking lactulose and/or protein supplementation (including taking glutamine) in the 4 weeks preceding the start of the study,
* Renal insufficiency (GFR<40mL/min), hepatic insufficiency (PT<70) or known heart disease,
* ATCD of digestive disease (celiac disease, chronic inflammatory bowel disease, abdominal surgery other than appendectomy or cholecystectomy),
* Occlusive or subocclusive syndrome,
* Digestive perforation or suspicion of perforation,
* Abdominal pain syndrome of undetermined cause,
* Chronic alcohol consumption (>14 units/week),
* Pregnant or parturient or breastfeeding woman or proven absence of contraception,
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/under guardianship or curatorship,
* Person participating in research participating in another trial / having participated in another trial within 2 weeks,
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or preventing them from giving informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the symptomatic effectiveness of glutamine supplementation in patients suffering from IBS-D with increased intestinal permeability | 8 weeks
  the change in Francis score measured before and after glutamine or placebo supplementation for 8 weeks in patients suffering from IBS-D with increased intestinal permeability.

IPD SHARING:
Plan to Share IPD: No